CLINICAL TRIAL: NCT05519241
Title: A Phase I Trial of Cancer-targeting Micelles for Non-myoinvasive Bladder Cancer
Brief Title: A Phase I Intravesical PPM Therapy for NMIBC
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ONCA-021-20S; VA Merit (Other Grant/Funding Number: 1I01CX002247)
Record Dates: First submitted 2022-08-18; First posted 2022-08-29 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Non-muscle-invasive Bladder Cancer
Keywords: non-muscle-invasive bladder cancer; BCG-refractory; paclitaxel; intravesical instillation
MeSH Terms: conditions — Non-Muscle Invasive Bladder Neoplasms

STUDY DESIGN:
Intervention Model Description: This is a Phase I, single-group, dose-escalation trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Phase I dose-escalation and expansion cohort (Experimental): There are three doses at the dose escalation stage: Dose level I: paclitaxel (PTX) 25 mg or 0.5 mg/ml; Dose Level II: PTX 50 mg or 1.0 mg/ml; Dose Level III: PTX 75 mg or 1.5 mg/ml. At the expansion cohort, up to 12 patients will be recruited and treated with PPM at the PTX dose of 50 mg or 1.0 mg/ml to determine the efficacy.
  Interventions: Drug: PLZ4-coated paclitaxel-loaded micelles (PPM)

INTERVENTIONS:
Drug: PLZ4-coated paclitaxel-loaded micelles (PPM) — PPM will be administrated weekly for 6 times through intravesical instillation into the bladder cavity

SUMMARY:
This clinical trial is to determine the safety and effectiveness of an investigational bladder cancer drug named "PLZ4-coated paclitaxel-loaded nanoscale micelle (PPM)." PPM is tiny particles that contain the chemotherapy drug paclitaxel. PLZ4 is a molecule that can possibly guide PPM to specifically target and deliver paclitaxel into and kill bladder cancer cells. In this trial, PPM will be instilled into the bladder cavity to treat bladder cancer that does not invade into the muscle layer of the bladder and that has failed the treatment of another drug BCG. Up to 29 patients will be enrolled into the trial. The main goal of this trial is to determine the dose of PPM for future clinical trials, assess the toxicity and obtain preliminary data regarding its effectiveness.

DETAILED DESCRIPTION:
The goal of this project is to conduct a Phase I clinical trial to determine the recommended Phase II dose (RP2D) of bladder cancer-targeting micelles loaded with a chemotherapeutic drug paclitaxel (PTX). The investigators previously developed a bladder cancer-specific targeting ligand named PLZ4, and a PLZ4-coated PTX-loaded nanoscale micelle (PPM) platform that can specifically deliver the drug load into bladder cancer cells both in vitro and in vivo. This proposed clinical trial is to conduct a first-in-human trial to use PPM for the treatment of non-myoinvasive bladder cancer (NMIBC). This primary objective of the proposed Phase I trial is to determine the recommended Phase II dose (RP2D) of PPM. The secondary objectives are to assess the toxicity, obtain preliminary efficacy information of PPM, and determine systemic absorption after intravesical instillation of PPM. Up to 29 patients with recurrent or refractory NMIBC after a standard first-line intravesical BCG treatment will be recruited. PPM will be given as intravesical instillation once weekly for six weeks. The toxicity will be assessed by the NCI Common Terminology Criteria for Adverse Events (CTCAE) version 5.0. The efficacy will be determined by urine cytology and cystoscopy after finishing treatment. Molecular correlative studies will be performed.

ELIGIBILITY:
Inclusion Criteria:

Patients must meet all of the following criteria to be eligible for study entry.

* Histologically confirmed bladder carcinoma in situ (CIS) urothelial or urothelial carcinoma, with or without T1 cancer. Patients are eligible if the biopsy was done within 3 months of enrollment and a cystoscopy demonstrates no gross disease invasion into muscularis propria within 4 weeks of enrollment.
* Patient must have BCG-unresponsive non-muscle-invasive bladder cancer (NMIBC) or intolerance of treatment with BCG. Treatment of pembrolizumab is not an inclusion or exclusion criteria as intravesical taxane probably has comparable efficacy as intravenous pembrolizumab. BCG-unresponsive disease is defined as being at least one of the following:

  * Persistent or recurrent CIS alone or with recurrent Ta/T1 (noninvasive papillary disease/tumor invades the subepithelial connective tissue) disease within 12 months of completion of adequate BCG therapy
  * Recurrent high-grade Ta/T1 disease within 6 months of completion of adequate BCG therapy
  * T1 high-grade disease at the first evaluation following an induction BCG course

In this context, adequate BCG therapy is defined as at least one of the following:

* At least five of six doses of an initial induction course plus at least two of three doses of maintenance therapy
* At least five of six doses of an initial induction course plus at least two of six doses of a second induction course

  * Refuse or intolerant of a radical cystectomy recommended by the treating urologist as the standard next therapy per urologic guidelines.
  * Age 18 years.
  * Performance status: ECOG performance status of 0, 1, or 2 (Appendix A) or Karnofsky performance status of 50 or higher (Appendix B).
  * Patient with life expectancy greater than 24 months.
  * No concurrent radiotherapy, chemotherapy, or other immunotherapy
  * No scheduled radiotherapy, chemotherapy, other immunotherapy, or surgery before the scheduled response evaluation.
  * Recovery from prior treatment side effects that might interfere with the study treatment, in the judgment of the participating urologist.
  * Laboratory tests performed within 14 days of study enrollment:
* Absolute neutrophil count (AGC/ANC) 1,500/uL
* Platelets 100,000/uL [Patients may be transfused to meet this requirement]
* Hemoglobin 8 g/dL [Patients may be transfused to meet this requirement]
* Calculated glomerular filtration rate (GFR) 50 mL/min/1.73m2
* Total bilirubin 2.0 X ULN (< 3 x ULN for patients with Gilbert's syndrome)
* AST, ALT, ALP 3.0 X ULN

  * Adequate pulmonary function with no clinical signs of severe pulmonary dysfunction.
  * Negative serum pregnancy test if the study participant is a female and of childbearing potential (non-childbearing is defined as greater than one year postmenopausal or surgically sterilized).
  * Female participants of childbearing potential must adhere to using a medically accepted method of birth control, i.e. a tubal ligation, an approved hormonal contraceptive or an intrauterine device, prior to screening and agree to continue its use during the study and up to 3 months after finishing this study or be surgically sterilized (e.g., hysterectomy or tubal ligation). Males must agree to use barrier methods of birth control while on study.
  * Provide signed informed consent and HIPAA authorization and agree to comply with all protocol-specified procedures and follow-up evaluations.

Exclusion Criteria:

Patients who meet any of the following criteria will be excluded from study entry.

* Existence of cancer at the upper urinary tract
* Concurrent use of other investigational agents.
* Evidence of regional and/or distant metastasis.
* NYHA (New York Heart Association) Class III or IV heart failure (Appendix C), uncontrollable supraventricular arrhythmias, any history of a ventricular arrhythmia, or other clinical signs of severe cardiac dysfunction.
* Symptomatic congestive heart failure (CHF), severe/unstable angina pectoris, or myocardial infarction within 6 months prior to study entry.
* Patient has an intractable bleeding disorder (e.g., coagulation factors deficiencies, Von Willebrand Disease).
* Patient taking medications that affect coagulation, such as aspirin (aspirin 81 mg oral once daily is allowed), Coumadin/Warfarin, heparin, low molecular weight heparin, direct thrombin inhibitors, and direct factor Xa inhibitors. Other nonsteroidal anti-inflammatory drugs (NSAIDs) are allowed as long as they are discontinued the day before therapy.
* History or evidence of uncontrollable central nervous system (CNS) disease.
* Active systemic infection requiring parenteral antibiotic therapy.
* Women who are pregnant or nursing.
* Psychiatric illness/social situations that would limit compliance with study requirements
* Other illness that in the opinion of the investigator would exclude the patient from participating in this study.
* Any other malignancy diagnosed within 3 years of trial entry with the exception of:

  * Basal or squamous cell skin cancers, or
  * Noninvasive cancer of the cervix, or
  * Any other cancer deemed to be of low-risk for progression or patient morbidity during trial period, such as localized prostate cancer after definitive treatment and prostate-specific antigen (PSA) less than 0.2 ng/ml.
* Patients unwilling to or unable to comply with the protocol.
* Patients with impaired decision-making capacity.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Estimated)
Dates: Start 2022-10-10 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
adverse events | up to 6 weeks after the last dose
  CTCAE v5.0 will be used to determine any adverse events and assess the grade. All toxicity as well as Grade 3 or higher adverse events will be analyzed.

SECONDARY OUTCOMES:
complete response rate | 6 weeks after finishing the last dose of PPM
  urine cytology, cystoscopy.

OTHER OUTCOMES:
blood paclitaxel concentration | within 6 hours after administration
  Blood will be drawn up to a few hours after the first dose of PPM at the expansion cohort to determine the systemic paclitaxel absorption.

CONTACTS AND LOCATIONS:
Overall Officials: Chong-Xian Pan, MD PhD, Principal Investigator — VA Boston Healthcare System Jamaica Plain Campus, Jamaica Plain, MA
Locations (1):
- VA Boston Healthcare System Jamaica Plain Campus, Jamaica Plain, MA, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
The published data is readily available after publications. Unpublished data will be available upon request. No individual participant data will be shared.